CLINICAL TRIAL: NCT06427330
Title: Phase II Study Assessing the Efficacy and Safety of Post-Transplant Low-Dose Inotuzumab Ozogamicin to Prevent Relapse of High Risk Acute Lymphoblastic Leukemia
Brief Title: Phase II Study of Post-Transplant Low-Dose Inotuzumab Ozogamicin to Prevent Relapse of Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IIT2024022
Record Dates: First submitted 2024-05-10; First posted 2024-05-23 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-04

CONDITIONS: Acute Lymphoid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inotuzumab ozogamicin (Experimental)
  Interventions: Drug: Inotuzumab ozogamicin

INTERVENTIONS:
Drug: Inotuzumab ozogamicin — 1. st dose is given after D+60：inotuzumab 0.3mg/m2
  2. nd dose is given after 1 month：inotuzumab 0.6mg/m2

SUMMARY:
To learn about the safety of post-HSCT two dose Inotuzumab Ozogamicin to participants with high risk B cell acute lymphoblastic leukemia(B-ALL). Also, to learn if giving Inotuzumab Ozogamicin to post-HSCT patients with high-risk B- ALL can help to reduce relapse and prolong disease free survival and overall survival.

DETAILED DESCRIPTION:
This is a Phase II study of inotuzumab ozogamicin for the treatment of patients who underwent transplantation for ALL and have a high risk of relapse. Participants will receive study treatment two doses until relapse of disease, unacceptable toxicity, or death, whichever occurs first Primary Objective

• To assess the efficacy of inotuzumab ozogamicin as measured by disease free survival (DFS) at one year.

Secondary Objective(s)

* To evaluate relapse rate, nonrelapse mortality (NRM), relapse, relapse-related mortality and overall survival (OS) at 1 year.
* To determine safety profile of inotuzumab ozogamicin after transplant including the incidence of hematological toxicity, secondary graft failure and other adverse event(AE)/severe adverse event(SAEs)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CD22-positive Acute Lymphoblastic Leukemia
* Patients who underwent an allogeneic hematopoietic stem cell transplantation(HSCT) from any donor source or auto-HSCT for acute lymphocytic leukemia
* Patients who are after T+60 after transplantation
* Patients who have/are either:

  * High risk B-ALL: (1) high white blood cell(WBC) count when newly diagnosed, (2) Poor risk group according to NCCN guideline 2021 of Acute Lymphoblastic
  * Leukemia
  * Relapsed or refractory to at least 1 line of treatment
  * Minimal residual disease(MRD) positive before HSCT, including flow cytometry and cytogenetic test
* Patients who have > 99% donor chimerism after allogeneic transplantation.
* Eastern Cooperative Oncology Group(ECOG) Performance status ≤ 2
* Participants must have ANC > 1,000/µL for 3 days and platelet transfusion independence as defined as a platelet count > 50,000/µL for 7 days.
* ≥ 18 years old, including male and female
* Participants must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with evidence of disease progression prior to enrollment
* Persistent prior treatment toxicities Grade 2 and above according to NCI CTCAE Version 4.03 (with the exception for alopecia, neuropathy, etc.)
* Patients with inadequate organ function and can't tolerate the study treatment determined by investigator as defined by:

  * Severe renal deficiency, with creatinine clearance < 50ml/min
  * Severe hepatic deficiency
  * Bilirubin, aspartate aminotransferase(AST), and/or ALT(ALT) > 2X institutional upper limit of normal
  * Severe cardiac or pulmonary deficiency
* Graft-versus-host disease(GVHD) grade III or IV (for patients with a prior allogeneic transplant).
* Active acute or chronic GVHD of the liver (for patients with a prior allogeneic transplant)
* History of veno-occlusive disease(VOD)
* Second active malignancy, other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast)
* Patients with uncontrolled inter-current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Serologic status reflecting active hepatitis B or C infection. Patients that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive patients will be excluded.)
* Any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the participant; or interfere with interpretation of study data.
* Known allergies, hypersensitivity, or intolerance to any of the study medications, excipients, or similar compounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
DFS | at one year after HSCT
  Efficacy as measured by DFS at one year, estimated using Kaplan-Meier, reported as median and 2-sided 80% and 95% Confidence Interval (CI) DFS is defined as "Time from date of HSCT to the date of disease progression (ie,objective progression, relapse from CR/CRi), or death due to any cause, whichever occurs first (including post-study treatment follow-up disease assessments)".

SECONDARY OUTCOMES:
Overall survival | at one year after HSCT
  Defined from time from HSCT to death due to any cause Defined from time from date of HSCT to death due to any cause, estimated using Kaplan-Meier, reported as median and 95% CI Difference in time-to-event endpoints will be tested using a 1-sided log-rank test at a significance level of 0.10
Relapse | at one year after HSCT
  Defined as time from date of HSCT to the date of first relapse. Reported as Cumulative Incidence
NRM | at one year after HSCT
  Defined as time from date of first dose to death due to any cause without prior relapse.
Incidence of hematological toxicity | at one year after HSCT
  Number of patients who develop hematological toxicity while on study, defined as grade of anemia, neutropenia and thrombocytopenia, etc.
Incidence of secondary graft failure(GF) | at one year after HSCT
  Number of patients who develop secondary graft failure while on study, defined as: Either cytopenias after initial engraftment (ANC <500/µL), with (a) donor chimerism of less than 5% or (b) falling donor chimerism with intervention such as second transplant or donor lymphocyte infusion (DLI) or (c) patient death due to cytopenias, and fall in donor chimerism, even if chimerism was >5%. Exclusion criteria for diagnosis of GF were (a) disease relapse (b) graft versus host disease or (c) other causes of cytopenias such as, viral infections, or drug induced
Percent of participants with AE/SAEs | at one year after HSCT
  safety profile of intervention as measured by percent of participants with any grade AE/SAEs

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, China